CLINICAL TRIAL: NCT06447181
Title: A Retrospective Cohort Study of Three- Dimensional Visualization Combined With ICG Molecular Fluorescence Imaging in Hepatolithiasis.
Brief Title: Application of Three- Dimensional Visualization Combined With ICG Molecular Fluorescence Imaging in Hepatolithiasis
Status: Not yet recruiting | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-KY-122-01
Record Dates: First submitted 2024-04-30; First posted 2024-06-07 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-04

CONDITIONS: Hepatolithiasis; Hepatectomy
Keywords: Three-dimensional visualization; ICG; hepatolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 3DVT-FI Group: Patients with hepatolithiasis using 3D visualization combined with ICG fluorescence technique
  Interventions: Device: 3D visualization technology ; ICG fluorescence technology .
- Conventional operation Group: Patients with hepatolithiasis using conventional operation

INTERVENTIONS:
Device: 3D visualization technology ; ICG fluorescence technology . — Three-dimensional reconstruction technology is a software that can collect CT and MRI data, perform image segmentation and three-dimensional reconstruction of the liver, gallbladder, dilated bile ducts, pancreas, venous, and arterial systems step by step.
  ICG fluorescence technology is a fluorescent laparoscopic technology that can detect extrahepatic biliary duct misalignment, improving surgical precision and safety.
  Groups: 3DVT-FI Group

SUMMARY:
This study adopted a retrospective study method to explore the clinical application value of 3D visualization combined with ICG molecular fluorescence imaging technology in hepatolithiasis, and further analyze whether 3D visualization combined with ICG molecular fluorescence imaging technology can improve the prognosis of hepatolithiasis by comparing with conventional surgery.

DETAILED DESCRIPTION:
Hepatolithiasis is a complex and intractable benign disease, often called "benign disease with poor prognosis". Clinical practice has proved that the diagnosis and treatment platform for hepatolithiasis built by modern digital image technologies such as 3D visualization and Indocine green fluorescence image navigation technology plays a vital leading role in accurate preoperative assessment, location of the lesion, formulation of the best surgical plan, and intraoperative navigation to avoid collateral damage. The clinical practice has proved that the diagnosis and treatment platform for hepatolithiasis built by modern digital image technologies such as 3D visualization and ICG fluorescence image navigation plays a vital leading role in accurate preoperative assessment, location of the lesion, formulation of the best surgical plan, and intraoperative navigation to avoid collateral damage.Therefore, we want to conduct a retrospective cohort study to explore the application value of 3D visualization combined with ICG fluorescence technology in hepatolithiasis, in order to further improve the curative effect of hepatolithiasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥18 years, of any gender; The diagnosis was hepatolithiasis；Surgical treatment has been performed.

Exclusion Criteria:

* Patients with severe cardiac, pulmonary, cerebral, renal dysfunction or other clinical contraindications who are unable to tolerate surgical treatment; Patients with malignant transformation; Lack of clinical data.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatolithiasis were ≥18 years old, and had undergone surgical treatment.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-08-30 (Estimated); Primary Completion 2024-12-25 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
operation time | Perioperative period
  minutes
intraoperative blood loss | Perioperative period
  ml
intraoperative incidental injuries | Perioperative period

SECONDARY OUTCOMES:
Postoperative complications | Perioperative period
  Bile leak, pancreatic leak and stone residue
Repeat surgery rate | Perioperative period
Serum bilirubin levels | Perioperative period
  mmol/L

CONTACTS AND LOCATIONS:
Locations (1):
- Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided